CLINICAL TRIAL: NCT07206004
Title: Effect of Parenteral Nutrition/Fluids on FibroScan Results in Patients With Short Bowel Syndrome
Brief Title: Effect of Parenteral Support on FibroScan in Short Bowel Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jessica Ramsing Wentworth, MD, Rigshospitalet, Denmark
Other Study IDs: H-25037724
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Short Bowel Syndrome; Intestinal Failure; Liver Diseases
Keywords: FibroScan; transient elastography; parenteral nutrition; intestinal failure; hepatic fibrosis
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure; Liver Diseases; Hyperphagia; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort - patients with short bowel syndrome on parenteral support: Patients will receive their ususal parenteral support during the study
  Interventions: Diagnostic Test: Fibroscan

INTERVENTIONS:
Diagnostic Test: Fibroscan — Fibroscan will be perfomed while the patient receives their usual parenteral support

SUMMARY:
Home Parenteral Support (HPS) is a life-sustaining treatment for patients with short bowel syndrome and intestinal failure. This study aims to investigate how administration of parenteral support affects FibroScan results in order to determine optimal timing of liver assessment in this patient population.

DETAILED DESCRIPTION:
The objective of this study is to investigate the applicability and accuracy of FibroScan in assessing liver status among patients with short bowel syndrome and intestinal failure, both before and after administration of PS, by assessing the immediate effect of PS administration on FibroScan results in patients with short bowel syndrome. This is of particular importance since the timing of FibroScan relative to PS administration and infusion volume is presumed to influence the results, and thereby potentially the interpretation of hepatic status.By understanding how parenteral support influences FibroScan measurements, we aim to optimize the use of this non-invasive technique for monitoring liver status in patients with intestinal failure, thereby defining the optimal timing of scanning in relation to PS administration. This could potentially enable earlier detection of hepatic complications and thereby improve the long-term prognosis for these patients.

Once included, participants must fast and abstain from fluids for 3 hours prior to the examination. Measurements will consist of a FibroScan, blood pressure, body weight, and bioimpedance analysis.

Measurements will be performed:

* Immediately before initiation of PS
* Two hours after initiation of PS
* Immediately after disconnection of PS
* Two hours after completion of PS Participants will collect urine from 0 to 14 hours. Spot urine sodium will be analyzed at 0 hours and 14 hours. Urine volume will be measured and then discarded. The standard infusion time for PS is set at 12 hours overnight.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with short bowel syndrome with capacity to give consent
* Patients receiving regular PS (≥4 days/week and ≥10 liters/week)
* Stable clinical condition

Exclusion Criteria:

* Known liver cirrhosis
* Active infection, severe dehydration, or electrolyte disturbances
* Pregnancy
* Receiving IV fluids or medications on study day
* Tapered infusion rate prior to disconnection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with short bowel syndrome receiving regular PS
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Fibroscran | 14 hours
  Change in transient elastography (FibroScan) values before, during, and after parenteral support

SECONDARY OUTCOMES:
CAP score | 14 hours
  Change in CAP score before, during, and after PS
Correlation of Fibroscan and PS | 14 hours
  Correlation of changes in FibroScan values with PS composition and volume
Correlation of Fibroscan and other factors | 14 hours
  Correlation with body weight, blood pressure, body fluid content, and urine output

CONTACTS AND LOCATIONS:
Overall Officials: Rahim M Naimi, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Digestive Diseases, Transplantation and General Surgery, Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pironi L, Sasdelli AS. Intestinal Failure-Associated Liver Disease. Clin Liver Dis. 2019 May;23(2):279-291. doi: 10.1016/j.cld.2018.12.009. Epub 2019 Feb 21. PMID 30947877
- [Background] de Ledinghen V, Vergniol J. Transient elastography (FibroScan). Gastroenterol Clin Biol. 2008 Sep;32(6 Suppl 1):58-67. doi: 10.1016/S0399-8320(08)73994-0. PMID 18973847
- [Background] Gu C, Wang H, Shu J, Zheng J, Li D, Cai C, Zhang P. RNA sequencing combining with whole exome sequencing reveals a compound heterozygous variant in ATM in a girl with atypical ataxia-telangiectasia. Clin Chim Acta. 2021 Dec;523:6-9. doi: 10.1016/j.cca.2021.08.026. Epub 2021 Aug 25. PMID 34453918
- [Background] Lee J, Lee R, Erpelding T, Siddoway RL, Gao J. The effect of water intake on ultrasound tissue characteristics and hemodynamics of adult livers. Clin Exp Hepatol. 2021 Jun;7(2):223-230. doi: 10.5114/ceh.2021.107068. Epub 2021 Jun 30. PMID 34295991
- [Background] Silva M, Costa Moreira P, Peixoto A, Santos AL, Lopes S, Goncalves R, Pereira P, Cardoso H, Macedo G. Effect of Meal Ingestion on Liver Stiffness and Controlled Attenuation Parameter. GE Port J Gastroenterol. 2019 Mar;26(2):99-104. doi: 10.1159/000488505. Epub 2018 Apr 20. PMID 30976614
- [Background] Alvarez D, Orozco F, Mella JM, Anders M, Antinucci F, Mastai R. Meal ingestion markedly increases liver stiffness suggesting the need for liver stiffness determination in fasting conditions. Gastroenterol Hepatol. 2015 Aug-Sep;38(7):431-5. doi: 10.1016/j.gastrohep.2015.01.009. Epub 2015 Mar 11. PMID 25769876
- [Background] Khunpakdee N, Jayanama K, Kaewdoung P, Promson K, Rattanasiri S, Warodomwichit D, Kantachuvesiri S, Sobhonslidsuk A. Transient Elastography in End-Stage Renal Disease Patients on Hemodialysis: The Effect of Net Fluid Withdrawal. Blood Purif. 2015;40(3):256-9. doi: 10.1159/000439582. Epub 2015 Oct 3. PMID 26430774
- [Background] Millonig G, Friedrich S, Adolf S, Fonouni H, Golriz M, Mehrabi A, Stiefel P, Poschl G, Buchler MW, Seitz HK, Mueller S. Liver stiffness is directly influenced by central venous pressure. J Hepatol. 2010 Feb;52(2):206-10. doi: 10.1016/j.jhep.2009.11.018. Epub 2009 Dec 4. PMID 20022130

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT07206004/Prot_SAP_000.pdf